CLINICAL TRIAL: NCT00133913
Title: Longitudinal Enumeration of Circulating Tumor Cells in Patients With Metastatic Colorectal Carcinomas
Brief Title: Circulating Tumor Cells in Patients With Metastatic Colorectal Cancer
Acronym: IMMC-06
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Immunicon (Industry)
Responsible Party: Senior Director, Clinical Development, Immunicon
Other Study IDs: IMMC-06
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2008-03-19 (Estimated); Status verified 2008-03

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients with measurable metastatic colorectal cancer about to start a new line of chemotherapy.
  Interventions: Procedure: Phlebotomy

INTERVENTIONS:
Procedure: Phlebotomy — Peripheral blood draws for testing of circulating tumor cells

SUMMARY:
This study enrolled patients with measurable metastatic colorectal cancer. Blood was drawn prior to the patient receiving a new therapy for his/her cancer and subsequently at 7-14 days, 3-4 weeks, and when an imaging study was done (~every 6 to 12 weeks). The blood was tested to find circulating tumor cells (CTCs) and to count them. The CTC levels were compared to the imaging study results to see if the CTC number and the imaging result (progression/no progression) were in agreement. Maximum active study participation was 12 months with up to 8 blood draws being taken. All patients are currently being followed for up to 24 months from their off study date for survival. The CTC result will also be used to see if there is a difference in survival and progression-free survival for those patients with and without a certain number of CTCs.

ELIGIBILITY:
Inclusion Criteria:

* Measurable metastatic carcinoma of the colon or rectum.
* 1st or 2nd line chemotherapy (3rd line acceptable with epidermal growth factor receptor [EGFR] targeted therapy)
* Chest/abdomen/pelvis scans every 6-12 weeks
* ECOG 0-2
* Hemoglobin (Hgb) > or = 8g/dl within 7 days prior to enrollment
* Age > or = to 18 years of age

Exclusion Criteria:

* Cumulative weekly blood draws exceeding 150mL/week
* Brain metastasis
* Prior history of other carcinoma within the last 5 years, except ductal carcinoma in situ (DCIS), non-invasive cervical cancer or non-melanoma skin cancer
* Surgery within 14 days of the initial blood draw, excluding surgical placement of a central venous device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology patients from academic institutions and private practices
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2004-03; Primary Completion 2007-01 (Actual); Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cohen, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Cohen SJ, Alpaugh RK, Gross S, O'Hara SM, Smirnov DA, Terstappen LW, Allard WJ, Bilbee M, Cheng JD, Hoffman JP, Lewis NL, Pellegrino A, Rogatko A, Sigurdson E, Wang H, Watson JC, Weiner LM, Meropol NJ. Isolation and characterization of circulating tumor cells in patients with metastatic colorectal cancer. Clin Colorectal Cancer. 2006 Jul;6(2):125-32. doi: 10.3816/CCC.2006.n.029. PMID 16945168
- [Derived] Coumans FA, Ligthart ST, Uhr JW, Terstappen LW. Challenges in the enumeration and phenotyping of CTC. Clin Cancer Res. 2012 Oct 15;18(20):5711-8. doi: 10.1158/1078-0432.CCR-12-1585. Epub 2012 Sep 25. PMID 23014524
- See also: 510(k) Premarket Notification — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfPMN/pmn.cfm?ID=25082